CLINICAL TRIAL: NCT01616992
Title: Interstitial Cystitis: Elucidation of the Psychophysiologic and Autonomic
Brief Title: Interstitial Cystitis: Elucidation of the Psychophysiologic and Autonomic Characteristics (ICEPAC) Study
Acronym: ICEPAC
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Thomas Chelimsky, Professor of Neurology, Case Western Reserve University
Other Study IDs: R01DK083538 (NIH)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Interstitial Cystitis/Painful Bladder Syndrome; Myofascial Pelvic Pain
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Interstitial Cystitis
  Interventions: Drug: Bupivacaine
- Myofascial Pelvic Pain
  Interventions: Drug: Bupivacaine
- Healthy
- First Degree Relative

INTERVENTIONS:
Drug: Bupivacaine — 20 ML dose of 0.75% Bupivacaine Instillation (into bladder) 1 time during second study visit.
  Groups: Interstitial Cystitis; Myofascial Pelvic Pain

SUMMARY:
Interstitial cystitis/painful bladder syndrome (IC/PBS) causes severe bladder pain and extensive disability in a large group of women int he prime of their productive lives. Extensive study of the bladder itself has uncovered many abnormalities, but the investigators do not know if these are the cause or result of the disorder. None of these has led to any real long-term progress in treatment, so far. The investigators have found that other autonomic disorders often occur in both the patients themselves and in the family members of patients with IC/PBS. The investigators therefore propose to determine whether the main abnormality in IC/PBS actually lies in the autonomic nervous system, rather than the bladder. The investigators will do this through careful measurements of autonomic function and sensation in patients who have IC/PBS, both at rest, and under controlled psychological stress. The investigators will compare their measurements to patients with myofascial pelvic pain, to know which abnormalities are truly linked to IC/PBS, and which simply reflect the presence of pelvic pain.

DETAILED DESCRIPTION:
The investigators primary hypothesis is that IC/PBS is a member of a larger family of disorders sharing aberrant central autonomic and sensory response to stress, pain or threat. These disorders appear to share a common vulnerability that seems to be conferred during development, and symptoms of these disorders usually are first manifested in response to an environmental trigger. This proposal aims to compare the neural, psychological, and endocrine phenotypes that characterize patients with IC/PBS with those of patients suffering myofascial pelvic pain (MPP) syndrome, an chronic pelvic pain distinct from IC/PBS, age-matched, healthy controls, and first degree relatives. These studies are designed to identify which levels of the neuraxis are impaired, both in the basal state, and in response to a well-characterized psychosocial stressor.

Aim 1: To differentiate the specific baseline neurophysiological abnormalities that occur in IC/PBS from those present in patients with MPP and healthy subjects, specifically:

1a: Bladder and pelvic floor afferent and efferent urogynecological function: (1) voiding diaries (efferent) modified to include void-state related numeric rating scales for pain (afferent); Uroflow measurements (efferent), and a double-blind placebo-controlled evaluation of the diagnostic lidocaine instillation test (afferent) with impact on voiding function (efferent); (2) semi-quantitative evaluation of pelvic floor function and identification of myofascial trigger points (efferent), including inter-observer validation of a standardized semi-quantitative examination (afferent); (3) quantitative Q-tip test for vulvodynia (afferent) (4) evaluation of dysmenorrhea (afferent) and menstrual function (efferent).

1b: somatic afferent and autonomic efferent neural function, specifically: (1) global screen for autonomic and neurological abnormalities through the established Small Fiber Score Instrument (SFIBS) questionnaire and structured neurological examination (afferent and efferent); (2) specific evaluation of sacral and lumbar nerve root function through a focused neurological examination (afferent and efferent); (3) parasympathetic cardiac function through the cardiac response to deep breathing (efferent); (4) sympathetic cardiac and vasomotor functions through the cardiovascular responses to the Valsalva maneuver and to an upright tilt table test (efferent); (5) sudomotor sympathetic function through the quantitative sudomotor axon reflex test (QSART) that evaluates post-ganglionic function (specifically abnormal in autonomic neuropathies) and through a thermoregulatory sweat test (efferent).

1. c: gastrointestinal afferent and efferent function, specifically upper bowel motility with established methods: (1) early satiety & gastric compliance by water load test (afferent). (2) gastric electrical activity through electrogastrography (efferent).

   Aim 2: To determine the specific developmental, psychiatric, pain, autonomic, and stress response characteristics common to IC/PBS and their family members, that differ from MPP and healthy subjects through:
2. a: Stress and trauma history in early childhood and adulthood.

2b: Psychiatric screening and psychometric quantitation of psychological symptoms, pain and function.

2c: Quantitation of associated co-morbid autonomic disorders through the ODYSA questionnaire.

2d: Salivary cortisol levels immediately prior to autonomic testing (anticipatory stress) and after a period of relaxation once the test is finished, in conjunction with a stress self-assessment inventory.

2e: Performance of the Trier test on a subset of patients and controls, with measurement of autonomic cardiovascular parameters, body temperature, catecholamine concentrations (norepinephrine, epinephrine, dopamine) and endocrine parameters: ACTH and adrenocortical hormones.

ELIGIBILITY:
General exclusion criteria for all IC/PBS and MPP patients, their siblings, and normal subjects will include presence of:

1. Currently attempting to become pregnant, pregnant (pregnancy test will be required) or breast feeding
2. Hematuria (? this can occur in IC) or infection on urinalysis
3. Recurrent urinary tract infections (> 3 culture documented episodes within the previous 12 months)
4. Pelvic or bladder neoplasm or infection
5. Inflammatory arthritis, connective tissue or auto-immune disorder
6. Evidence of unstable medical disorder, such as kidney (rising creatinine, or end-stage renal failure) or liver impairment (rising AST or ALT, or end-stage with coagulopathy), poorly controlled significant cardiovascular (CHF), respiratory, endocrine (diabetes - A1c > 9 - or untreated thyroid dysfunction) or uncontrolled psychiatric illness (such as untreated depression, psychosis, etc.).
7. Neuropathy, central nervous system disorder (e.g., Parkinson's Disease, Alzheimer's, MS, stroke, etc)
8. Treatment with a drug or medical device within the previous 30 days that has not received regulatory approval
9. Use of hormones (except insulin, thyroid replacement or oral contraceptives, which will be carefully documented)
10. Regular use of opiods
11. Allergy to lidocaine
12. Inability to stop use of autonomically active or pro-kinetic (gastrointestinal motility modifying) agents for a minimum of 5 half-lives prior to testing
13. Current substance abuse or > 10 alcoholic beverages per week
14. Any major surgical intervention with general anesthesia in the last 90 days
15. Any on-going or pending medical, health or disability related litigation, or current pursuit of disability
16. Any condition that in the judgment of the investigator and the internal advisory panel would interfere with the patient's ability to provide informed consent, comply with study instructions, place the patient at increased risk, or which would clearly confound the interpretation of the study results (specific reason will be documented) 17.Investigators, study staff and their immediate families 18.Inability to speak English

19) Previously completed or withdrawn from this study

Normal controls and siblings: Aged-matched healthy female subjects will be recruited by nomination by patients and advertisement. A history and physical will be obtained by a physician, and controls will be required to have no history, symptoms or signs of (exclusion criteria):

1. FM or CFS (unexplained fatigue for a period of 6 months or more)
2. IC/PBS, MPP or chronic pelvic discomfort or chronic pain disorder of any type.
3. One of the other ODYSA dysautonomias

IC/PBS Patients - The diagnosis of IC/PBS will be made using most current NIDDK criteria. Exclusion criteria:

1. Intravesical therapy or bladder hydrodistention within the previous 90 days
2. Initiation of pentosan polysulfate sodium (Elmiron) within the previous 90 days
3. Previous augmentation cystoplasty, cystectomy or cytolysis, neurectomy (i.e., hypogastric nerve plexus ablation) or implanted neural stimulator which is functionally "on", in active use, or unable to be turned functionally off throughout the study period.

MPP Patients - Inclusion Criteria

1. CPP > 3 months duration, with pain ranked > 3/10 by oral analog scale
2. Presence of 1 or more palpable trigger points on transvaginal and/or transrectal examination of the pelvic floor, which reproduces the pain for which they are seeking medical care.

Exclusion criteria:

1. Pelvic surgery within the last 12 months
2. Pelvic injection with the last 90 days
3. Presence of IC/PBS by the current NIDDK criteria

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population will be composed of four subject groups:
  Group I: This group will consist of female IC/PBS patients (n = 76) Group II: This group will consist of female siblings of patients (n = 38) Group III: This group will consist of female MPP patients (n = 76) Group IV: This group will consist of healthy female control subjects (n = 38) Female subjects ages 18-80 will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Interstitial Cystitis | 1 month
  Clinical Assessment
Myofascial Pelvic Pain | 1 Month
  Clinical Assessment

SECONDARY OUTCOMES:
Depression Symptoms | 1 Month
  Questionnaire Assessment of Symptoms
Stress Symptoms | 1 month
  Questionnaire Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Chelimsky, MD, Principal Investigator — Medical College of Wisconsin; Jeffrey Janata, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - Summa Health System, Akron, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio

REFERENCES:
- [Derived] Williams DP, Chelimsky G, McCabe NP, Koenig J, Singh P, Janata J, Thayer JF, Buffington CA, Chelimsky T. Effects of Chronic Pelvic Pain on Heart Rate Variability in Women. J Urol. 2015 Nov;194(5):1289-94. doi: 10.1016/j.juro.2015.04.101. Epub 2015 May 9. PMID 25963185